CLINICAL TRIAL: NCT06710964
Title: Inducing Self-Dehumanization to Examine the Effects on Oxytocin and Suicide Risk
Brief Title: Inducing Self-Dehumanization to Examine Oxytocin and Suicide Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Thomas Joiner, Robert O. Lawton Distinguished Professor of Psychology, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FP00007283
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Mechanistic Self-Dehumanization Condition; Control Condition
Keywords: self-dehumanization; suicidal ideation; oxytocin
MeSH Terms: conditions — Suicidal Ideation | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mechanistic Self-Dehumanization Condition (Experimental): A self-dehumanized future condition (i.e., a futuristic paradigm that likens the individual to a machine)
  Interventions: Other: The Ten Item Personality Inventory; Other: Mechanistic Self-Dehumanization Condition; Other: Debrief; Diagnostic Test: Clinical Interview; Other: Self-Report Measures; Other: Blood Draw
- Control Condition (Active Comparator): Control Condition
  Interventions: Other: The Ten Item Personality Inventory; Other: Control Condition; Diagnostic Test: Clinical Interview; Other: Self-Report Measures; Other: Blood Draw

INTERVENTIONS:
Other: The Ten Item Personality Inventory — The Ten Item Personality Inventory (TIPI) is a brief self-report measure of the Big Five personality dimensions, which will provide the mock basis for the self-dehumanization induction. Participants will indicate responses on 7-point Likert scale ranging from 1 ("disagree strongly") to 7 ("agree strongly").
  Building off previously validated tasks participants will be told that the TIPI measure provided certain information about their personalities (and therefore expectations for their future). To establish credibility, participants will receive accurate feedback surrounding their reported levels of extraversion (high, medium, low). Participants will be randomly assigned to receive one of the following pre-written, feedback scripts as additional implications about their extraversion scores in relationship to future social expectations.
Other: Mechanistic Self-Dehumanization Condition — Future Mechanistic Self-Dehumanization Script: "Based on your responses, you're the type who will feel at times that you're just a number in the system. The day-to-day pattern of going to work and fulfilling responsibilities will seem repetitive, like you are a mechanical device just going through the motions. You might find that relationships feel distant or lack the warmth you seek, making it challenging to form deeper connections. Over time, each day will blend into the next, which will likely lead to you operating on autopilot, existing among humans."
  Arms: Mechanistic Self-Dehumanization Condition
Other: Debrief — Debrief: Those in the self-dehumanized condition will receive a brief rehumanization intervention to undo the effects of the self-dehumanized condition. This intervention will involve a reminder that the condition was fabricated and will involve reading quotes involving general themes of humanness. The participants will then share with the experimenter how they connect to their humanness. The experimenter will document responses and encourage engagement in humanizing activities following the study visit. Findings from these qualitative responses will inform a rehumanization intervention in another study.
  Arms: Mechanistic Self-Dehumanization Condition
Other: Control Condition — Future Control Script: "Based on your responses, you're the type who will have a very normal life. You will wake up, go to your job during the weekdays, and complete all necessary tasks. On the weekends you will spend time doing fulfilling activities. Relationships will have natural ups and down, but overall, you will feel satisfied by your connectedness to others. Though some days may feel monotonous, you will feel relaxed knowing you belong."
  Arms: Control Condition
Diagnostic Test: Clinical Interview — Clinical Interview. Self-Injurious Thoughts and Behaviors Interview-Short Form (SITBI-SF). Participants will complete an in-person interview featuring 72-items about their history of self-injury and suicidal behaviors. This interview includes 6 yes/no style questions about suicidal thoughts, suicidal plans, suicidal gestures, suicidal attempts, nonsuicidal self-injury thoughts, and nonsuicidal self-injury. Each category that is endorsed, across the lifetime, has follow up questions surrounding times, duration, intensity, severity, type, and if medical attention was sought. This interview has sound psychometric properties.
Other: Self-Report Measures — Depressive Symptom Index - Suicidality Subscale (DSI-SS). Patient Health Questionnaire-8 (PHQ-8). Interpersonal Needs Questionnaire (INQ). Self-Dehumanization Scale (SDS).
Other: Blood Draw — Five milliliters of blood will be drawn before and after study interventions for the quantification of plasma oxytocin concentrations by certified phlebotomists. Samples will be collected into chilled Ethylenediaminetetraacetic Acid (EDTA) tubes, inverted ten times to mix with anticoagulants, and centrifuged at 1600g for 15 minutes at 4˚C. Cleared plasma will be aliquoted into cryotubes and stored at -80˚C. Consistent with expert recommendations, oxytocin levels will be obtained from the samples diluted 1:4 (i.e., oxytocin can be discarded through plasma proteins when incorporating an extraction step before conducting the enzyme-linked immunosorbent assay [ELISA]). Second, to buffer against contrasting concerns, an aliquot of each sample will be analyzed for test-retest purposes. Oxytocin concentrations will be measured using a validated commercially available and sensitive ELISA neurophysin kit (Abcam).

SUMMARY:
The goal of this experiment is to further determine if self-dehumanization is a novel risk factor for suicide. This study will induce self-dehumanization using a novel experimental self-dehumanized future condition (i.e., a futuristic paradigm that likens the individual to a machine) and compare this group to a control group to analyze the pathway between higher perceptions of self-dehumanization, suicidal ideation, and changes in oxytocin concentrations.

It is hypothesized that participants randomly assigned to the self-dehumanized mechanistic future condition will exhibit temporary increases in suicidal ideation (which will be thoroughly assessed, intervened upon following the induction) and decreases in oxytocin concentrations as compared to the control condition, which will not display significant changes. Further, we will explore if the magnitude of the oxytocin response will partially mediate the change in suicidal ideation.

DETAILED DESCRIPTION:
Purpose: Humans are inherently social beings, and the need for belonging and connection is fundamental. Severe perceptions of social exclusion, non-belonging, and isolation can result in significant psychological harm, including suicide, which claims nearly 50,000 lives annually in the U.S. and affects over 13 million individuals through suicidal ideation (SI). A key predictor of SI, thwarted belongingness, arises from feelings of exclusion and non-belonging, yet more specificity is needed to identify the types of non-belonging that contribute most to suicide risk. Self-dehumanization-a perception of oneself as less than human-emerges as a promising factor in understanding and mitigating SI, with empirical evidence linking it to anxiety, depression, suicidal ideation, and social withdrawal. Preliminary research suggests that self-dehumanization is influenced by neurobiological processes, particularly oxytocin, a hormone critical to social connectedness and self-perception. Low oxytocin levels have been linked to self-dehumanization, reduced social reengagement, and heightened suicide risk, highlighting its potential as a target for intervention. Building on these insights, this study will experimentally induce and reduce self-dehumanization to examine its effects on SI and oxytocin levels. Thus, this study will use a self-dehumanization induction to analyze its impact on SI and oxytocin. Findings will provide a novel framework for integrating psychotherapeutic and neurobiological strategies into suicide prevention efforts.

Research Design/Method: The present study will utilize an experimental design with two groups, an experimental self-dehumanization induction group and a comparison control group.

Procedure: All interested participants will be instructed to fill out the screening survey to determine fit. Eligible participants will be invited to complete the study visit in person. Following consent, participants will complete a pre-induction fasted blood draw of 5 milliliters (i.e., approximately a tablespoon of blood). Next, participants will complete the Self-Injurious Thoughts and Behaviors-Short Form interview with the experimenter and a battery of randomized self-report assessments. After completion, participants will fill out a personality inventory distractor. Eligible participants will then be randomly assigned to one of two experimental conditions and provided a futuristic report based upon the false reports of the personality inventory. The two conditions will either be the mechanistic self-dehumanization condition or the control condition. Following this, they will undergo a post-induction 5 milliliter fasted blood draw. They will then complete a post-induction battery of self-report measures. Participants will be queried for any changes in suicide risk and any current suicidal ideation and intent will receive appropriate interventions (e.g., means safety counseling, safety planning). Upon completion participants will be debriefed, provided a brief rehumanization remedy to undo the effects of the self-dehumanized condition, compensated, and provided mental health resources (e.g., the National Suicide Prevention Lifeline). The appointment is expected to take approximately 1.5 hours to complete

Data Analyses: All results will be analyzed in R. First, descriptive statistics and zero-order bivariate correlation analyses will be assessed. For Study 1, repeated measures ANCOVAs will be used to examine group differences (i.e., the active self-dehumanization condition and control condition) in changes in oxytocin levels, self-dehumanization scores, and suicidal ideation, controlling for social isolation (i.e., thwarted belongingness, a factor of the Interpersonal Needs Questionnaire). Post-hoc pairwise comparisons will be conducted if the omnibus test indicates statistically significant effects. Following this, exploratory analyses will be conducted to assess if oxytocin partially mediates the relationship between self-dehumanization pre-experimental manipulation and suicide risk post-experimental manipulation (controlling for suicide risk at pre-experimental manipulation) through bootstrapped mediation procedures (i.e., 10,000 samples using the mediation and lavaan packages in R).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 40
* Biological females will be screened to ensure that they have a regular menstrual cycle with a length of 26-30 days and will be scheduled according to their cycle (see Research Strategy for details).
* At least a moderate level of self-dehumanization (i.e., a sum score of 12 or greater out of a possible score of 28) and lifetime suicidal ideation

Exclusion Criteria:

* A phobia of needles (i.e., Trypanophobia)
* Any medical conditions precluding them from engaging in a 10-hour fast (consumption of water is allowed and encouraged)
* Life-threatening suicide risk which would result in taking appropriate steps to ensure safety of the individual (e.g., hospitalization)
* A psychosis-related diagnosis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change in Suicidal Ideation | Baseline and 1 hour later after the experimental induction
  Suicidal Ideation will be measured using the Depressive Symptom Index-Suicidality Subscale (DSI-SS) where the scores range from 0-12 and higher scores indicate higher levels of suicidal ideation. These analyses will control for Baseline suicidal ideation and the thwarted belongingness sub-scale from the Interpersonal Needs Questionnaire where thwarted belongingness scores range from 1-56 and higher scores indicate greater perceptions of thwarted belongingness.
Change in Oxytocin Levels | Baseline and 1 hour later after the experimental induction
  Five milliliters of blood will be drawn before and after study interventions for the quantification of plasma oxytocin concentrations by certified phlebotomists (including the PI, who is already certified and currently collecting samples for a T-32 supported project). Samples will be collected into chilled EDTA tubes, inverted ten times to mix with anticoagulants, and centrifuged at 1600g for 15 minutes at 4˚C. Cleared plasma will be aliquoted into cryotubes and stored at -80˚C. Consistent with expert recommendations, oxytocin levels will be obtained from the samples diluted 1:4 (i.e., oxytocin can be discarded through plasma proteins when incorporating an extraction step before conducting the enzyme-linked immunosorbent assay [ELISA]). Second, to buffer against contrasting concerns, an aliquot of each sample will be analyzed for test-retest purposes. Oxytocin concentrations will be measured using a validated commercially available and sensitive ELISA neurophysin kit (Abcam).

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol will be designed to allow for IPD sharing. IPD de-identified demographic, self-report, and neurobiological (i.e., oxytocin) data may be shared. Data will not be shared if the participant denies to share their data. Data will be accessible by contacting the Central Contact Person of the study: Morgan Robison (mrobison@psy.fsu.edu). If data are uploaded to a public repository, the external link will be made available here.

REFERENCES:
- [Background] Robison M, Abderhalden FP, Joiner TE. Dehumanization and the Association With Nonsuicidal Self-Injury and Suicidal Ideation in an Incarcerated Population. Crisis. 2024 Jul;45(4):287-293. doi: 10.1027/0227-5910/a000952. Epub 2024 Mar 5. PMID 38441129
- [Background] Robison M, Jeon ME, Udupa NS, Potter M, Robertson L, Joiner T. The Self-Dehumanization Scale: Three Studies on Its Development and Validation. J Pers Assess. 2025 Jan-Feb;107(1):41-57. doi: 10.1080/00223891.2024.2367543. Epub 2024 Jun 28. PMID 38940620